CLINICAL TRIAL: NCT02963922
Title: Effect and Safety of Liraglutide 3.0 mg in Subjects With Overweight or Obesity and Type 2 Diabetes Mellitus Treated With Basal Insulin
Acronym: SCALE™ Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4272; U1111-1177-4903 (Other: World Health Organization (WHO)); 2015-005619-33 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- liraglutide 3.0 mg (Experimental)
  Interventions: Drug: Liraglutide 3.0 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide 3.0 mg — Injected subcutaneously (s.c., under the skin) once daily
  Arms: liraglutide 3.0 mg
Drug: Placebo — Injected subcutaneously (s.c., under the skin) once daily
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate effect and safety of liraglutide 3.0 mg in subjects with overweight or obesity and type 2 diabetes mellitus treated with basal insulin.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Diagnosed with type 2 diabetes mellitus - Treatment with up to 2 OADs (oral anti-diabetic) (metformin, glitazone, SGLT-2 inhibitor (sodium-glucose cotransporter-2 inhibitors) or sulphonylurea) - Stable treatment with basal insulin according to its label (no requirement of minimum or maximum dose) for at least 90 days prior to screening, as judged by the investigator - HbA1c (glycosylated haemoglobin) 6.0-10.0% (both inclusive) - BMI (body mass index) equal to or above 27 kg/m^2 - Age at least 18 years at the time of signing informed consent Exclusion Criteria: - Diagnosis of type 1 diabetes - Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8 (see Section 8.2.3) - Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator - Unable or unwilling to perform self-monitoring of plasma glucose according to the protocol and to keep a diabetes diary - Treatment with any hypoglycaemic medications other than OADs and basal insulin within the past 90 days prior to screening - Treatment with a DPP-IV (dipeptidyl peptidase-4) inhibitor within the past 90 days prior to screening - Recent history of cardiovascular disease (myocardial infarction or stroke within the past 6 months), severe congestive heart failure (NYHA class III, IV), or second degree or greater heart block - Personal or family history of Medullary Thyroid Carcinoma (MTC) or Multiple Endocrine Neoplasia type 2 (MEN2) - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) - For Germany: Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine device), or sexual abstinence or vasectomised partner - Use in past 90 days of medications known to induce significant weight loss (e.g., prescription weight loss medications) or weight gain (e.g., chronic use of oral steroids, second generation antipsychotics) - History of pancreatitis (acute or chronic) - History of major depressive disorder within the past 2 years - Any lifetime history of a suicide attempt - Inadequately treated blood pressure defined as Grade 3 hypertension or higher (Systolic above or equal to 180 mmHg or diastolic above or equal to110 mmHg). - History of malignancy (except for non-melanoma skin cancer) within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (17):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Winchester, Virginia
- Canada (8):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
  - Novo Nordisk Investigational Site, Québec
- Germany (8):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (4):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Rome
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Garvey WT, Birkenfeld AL, Dicker D, Mingrone G, Pedersen SD, Satylganova A, Skovgaard D, Sugimoto D, Jensen C, Mosenzon O. Efficacy and Safety of Liraglutide 3.0 mg in Individuals With Overweight or Obesity and Type 2 Diabetes Treated With Basal Insulin: The SCALE Insulin Randomized Controlled Trial. Diabetes Care. 2020 May;43(5):1085-1093. doi: 10.2337/dc19-1745. Epub 2020 Mar 5. PMID 32139381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 53 sites in Canada (7), Germany (7), Israel (6), Italy (4), Mexico (2), Turkey (7) and United States (20).
Pre-assignment Details: Participants were randomised in a 1:1 manner to receive either liraglutide or placebo as an adjunct to a reduced-calorie diet and increased physical activity as part of a comprehensive lifestyle intervention program.
Groups:
- Liraglutide 3.0 mg: Participants received liraglutide once daily by subcutaneous injection irrespective of the timing of meals. Participants received 0.6 milligrams (mg) liraglutide during the first week. The dose was escalated in weekly increments of 0.6 mg until the maintenance dose of 3.0 mg was reached after 4 weeks. The treatment period was 56 weeks.
- Placebo: Participants received matching placebo once daily by subcutaneous injection irrespective of the timing of meals. Dose escalation for placebo matched that of liraglutide. The treatment period was 56 weeks.
Period: Overall Study
Arm/Group | Liraglutide 3.0 mg | Placebo
Started | 198 | 198
Completed | 166 | 168
Not Completed | 32 | 30
Not completed — Adverse Event | 15 | 6
Not completed — Protocol deviation | 6 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Other | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Liraglutide 3.0 mg: Participants received liraglutide once daily by subcutaneous injection irrespective of the timing of meals. Participants received 0.6 mg liraglutide during the first week. The dose was escalated in weekly increments of 0.6 mg until the maintenance dose of 3.0 mg was reached after 4 weeks. The treatment period was 56 weeks.
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 198 | 198 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.3) | 57.6 (10.4) | 56.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 99 | 207
  Male | 90 | 99 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 29 | 72
  Not Hispanic or Latino | 155 | 169 | 324
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race is presented.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 3 | 5 | 8
    Black or African American | 17 | 11 | 28
    Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    White | 174 | 180 | 354
    Other | 0 | 2 | 2
Body weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 100.6 (20.8) | 98.9 (19.9) | 99.7 (20.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Change in body weight from baseline (week 0) to week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for adverse events [AEs]) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage change
  In-trial observation period: number analyzed (Participants) | 191 | 193
  In-trial observation period | -6.0 (6.0) | -1.5 (5.4)
  On-drug observation period: number analyzed (Participants) | 163 | 168
  On-drug observation period | -6.5 (5.8) | -1.7 (5.2)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach. Week 56 responses were analysed using an analysis of covariance model with treatment, body mass index (BMI) groups and sex as factors and baseline body weight as covariate; Test type: Superiority — The treatment policy estimand evaluated the treatment effect (liraglutide 3.0 mg vs placebo) at week 56 for all randomised participants regardless of premature discontinuation of trial product; p < .0001, ANCOVA; Treatment difference = -4.32, 95% CI 2-sided [-5.48 to -3.16], Standard Error of Mean 0.59 — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of on-drug before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups and sex as factors and baseline body weight as covariate, all nested within visit; Test type: Superiority — The hypothetical estimand evaluated the treatment effect (liraglutide 3.0 mg vs placebo) for all randomised participants assuming that all participants remained on trial product (on-treatment principle); p < .0001, MMRM; Treatment difference = -5.10, 95% CI 2-sided [-6.30 to -3.91], Standard Error of Mean 0.61 — Liraglutide 3.0 mg - placebo

2. Primary Outcome: Participants Losing at Least 5% of Baseline Body Weight
Description: The estimated percentage of participants losing at least 5% of baseline (week 0) body weight at week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for adverse events [AEs]) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants
  In-trial observation period: number analyzed (Participants) | 191 | 193
  In-trial observation period | 51.80 | 23.98
  On-drug observation period: number analyzed (Participants) | 195 | 197
  On-drug observation period | 56.92 | 21.83
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach. Week 56 responses were analysed using a logistic regression model with treatment, BMI groups and sex as factors and baseline body weight as covariate; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.41, 95% CI 2-sided [2.19 to 5.31] — Liraglutide 3.0 mg/Placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of on-drug before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups and sex as factors and baseline body weight as covariate, all nested within visit. The MMRM was used to classify responders and analysed with a logistic regression with treatment as the only factor; Test type: Superiority; p < .0001, Mixed model for repeated measurements; Odds Ratio (OR) = 4.73, 95% CI 2-sided [3.04 to 7.36] — Liraglutide 3.0 mg/Placebo

3. Secondary Outcome: Participants Losing More Than 10% of Baseline Body Weight at Week 56
Description: The estimated percentage of participants losing more than 10% of baseline (week 0) body weight at week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for adverse events [AEs]) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants
  In-trial observation period: number analyzed (Participants) | 191 | 193
  In-trial observation period | 22.77 | 6.55
  On-drug observation period: number analyzed (Participants) | 195 | 197
  On-drug observation period | 22.56 | 5.58

4. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for AEs) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Centimeters (cm)
  In-trial observation period: number analyzed (Participants) | 189 | 193
  In-trial observation period | -5.40 (6.06) | -2.60 (5.72)
  On-drug observation period: number analyzed (Participants) | 163 | 168
  On-drug observation period | -5.71 (6.05) | -2.78 (5.63)

5. Secondary Outcome: Change in HbA1c
Description: Change in glycosylated haemoglobin (HbA1c) from baseline (week 0) to week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for AEs) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of HbA1c
  In-trial observation period: number analyzed (Participants) | 187 | 188
  In-trial observation period | -1.1 (1.2) | -0.5 (1.2)
  On-drug observation period: number analyzed (Participants) | 160 | 164
  On-drug observation period | -1.2 (1.1) | -0.7 (1.0)

6. Secondary Outcome: Change in FPG
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to week 56 was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for AEs) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Millimoles per liter (mmol/L)
  In-trial observation period: number analyzed (Participants) | 187 | 188
  In-trial observation period | -0.91 (3.13) | -0.68 (3.04)
  On-drug observation period: number analyzed (Participants) | 162 | 165
  On-drug observation period | -1.05 (3.08) | -0.96 (2.68)

7. Secondary Outcome: Change in Short Form-36 (SF-36) v2.0 Acute, Physical Functioning Score
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline (week 0) in SF-36 physical functioning score was presented based on in-trial data and on-drug data. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale
  In-trial observation period: number analyzed (Participants) | 186 | 187
  In-trial observation period | 2.5 (7.9) | 2.6 (7.3)
  On-drug observation period: number analyzed (Participants) | 161 | 167
  On-drug observation period | 2.9 (7.8) | 2.5 (7.1)

8. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT), Physical Function Domain (5-items) Score
Description: Change in IWQoL-Lite for CT physical function domain (5-items) score. IWQoL-Lite for CT is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. The endpoint was presented based on in-trial data and on-drug data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which participants are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for AEs) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale
  In-trial observation period: number analyzed (Participants) | 186 | 187
  In-trial observation period | 7.3 (22.5) | 6.8 (21.5)
  On-drug observation period: number analyzed (Participants) | 161 | 167
  On-drug observation period | 8.2 (20.9) | 6.5 (21.8)

9. Secondary Outcome: Change in Total Daily Insulin Dose (U)
Description: Change in total daily insulin dose from baseline (week 0) to week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Units of insulin dose (U)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Units of insulin dose (U) | 3 (30) | 18 (38)

10. Secondary Outcome: Change in Total Daily Basal Insulin Dose (% of Pre-trial Dose in U)
Description: Change in total daily basal insulin dose from baseline (week 0) to week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage change | 19 (121) | 64 (139)

11. Secondary Outcome: Change in Total Daily Basal Insulin Dose (U/kg)
Description: as for outcome 10
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Units of insulin dose per kilogram(U/kg)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Units of insulin dose per kilogram(U/kg) | 0.05 (0.33) | 0.15 (0.30)

12. Secondary Outcome: Change in Total Daily Insulin Dose (U/kg)
Description: as for outcome 9
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
U/kg | 0.05 (0.33) | 0.18 (0.37)

13. Secondary Outcome: Change in 7-point SMPG Profile Mean Daytime Glucose Value
Description: Participants measured plasma glucose values using the blood glucose meter at 7 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner and at bedtime. Change from baseline (week 0) to week 56 in 7-point self-measured plasma glucose (SMPG) profile mean daytime glucose value was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
mmol/L | -2.2 (2.6) | -1.6 (2.8)

14. Secondary Outcome: Change in sBP and dBP
Description: Change in systolic blood pressure (sBP) and diastolic blood pressure (dBP) from baseline (week 0) to week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Millimeters of mercury (mmHg)
  sBP: number analyzed (Participants) | 188 | 192
  sBP | -6 (14) | -2 (15)
  dBP: number analyzed (Participants) | 188 | 192
  dBP | -3 (9) | -1 (9)

15. Secondary Outcome: Change in Lipids -Total Cholesterol, HDL, LDL, VLDL, Triglycerides and FFA
Description: Change in total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, very low density lipoprotein (VLDL) cholesterol, triglycerides and free fatty acids (FFA) from baseline (week 0) to week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
mmol/L
  Total cholesterol: number analyzed (Participants) | 186 | 190
  Total cholesterol | -0.12 (0.82) | 0.04 (0.69)
  HDL cholesterol: number analyzed (Participants) | 186 | 190
  HDL cholesterol | 0.05 (0.17) | 0.03 (0.17)
  LDL cholesterol: number analyzed (Participants) | 186 | 190
  LDL cholesterol | -0.08 (0.72) | 0.05 (0.57)
  VLDL cholesterol: number analyzed (Participants) | 186 | 190
  VLDL cholesterol | -0.09 (0.35) | -0.04 (0.33)
  Triglycerides: number analyzed (Participants) | 186 | 190
  Triglycerides | -0.21 (0.89) | -0.08 (0.80)
  Free fatty acids: number analyzed (Participants) | 182 | 188
  Free fatty acids | -0.10 (0.27) | -0.06 (0.34)

16. Secondary Outcome: Change in SF-36: Sub-domains
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in the sub-domain scores was presented based on in-trial data. A positive change score indicates an improvement since baseline. Results are presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale
  Bodily Pain: number analyzed (Participants) | 186 | 187
  Bodily Pain | 1.2 (8.3) | 1.2 (9.1)
  General Health: number analyzed (Participants) | 186 | 187
  General Health | 1.9 (7.8) | 0.3 (7.7)
  Physical Functioning | 2.5 (7.9) | 2.6 (7.3)
  Role-physical: number analyzed (Participants) | 186 | 187
  Role-physical | 0.8 (7.7) | 0.9 (8.0)
  Role Lim Emotion Prob: number analyzed (Participants) | 186 | 187
  Role Lim Emotion Prob | -1.2 (8.1) | -0.3 (8.2)
  Mental Health: number analyzed (Participants) | 186 | 187
  Mental Health | -1.1 (8.6) | -1.1 (7.5)
  Social Functioning: number analyzed (Participants) | 186 | 187
  Social Functioning | -0.7 (7.7) | -0.6 (6.3)
  Vitality: number analyzed (Participants) | 186 | 187
  Vitality | 1.0 (8.0) | -0.0 (7.7)

17. Secondary Outcome: Change in SF-36: Physical Component Summary (PCS)
Description: Change in short form 36 v2.0 acute domain physical component summary (PCS) from baseline (week 0) to week 56 was presented based on in-trial data. SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. It consists of 2 component summary measures that further summarize 8 health domain scales. The physical component summary (PCS) measure is derived from domain scales of physical functioning, role-physical, bodily pain, and general health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale | 2.7 (7.5) | 2.2 (7.2)

18. Secondary Outcome: Change in SF-36: Mental Component Summary (MCS)
Description: Change in short form 36 v2.0 acute domain mental component summary (MCS) from baseline (week 0) to week 56 was presented based on in-trial data. SF- 36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The mental component summary (MCS) measure is derived from domain scales of vitality, social functioning, role emotional and mental health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale | -1.9 (7.9) | -1.7 (6.8)

19. Secondary Outcome: Change in IWQoL-Lite for CT: Pain/Discomfort Domain Score
Description: Change in IWQoL-Lite for CT pain and discomfort domain from baseline (week 0) to week 56 was presented based on in-trial data. IWQoL-Lite for CT is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale | 4.0 (22.1) | 4.6 (23.1)

20. Secondary Outcome: Change in IWQoL-Lite for CT: Psychosocial Domain Score
Description: Change in IWQoL-Lite for CT psychosocial domain from baseline (week 0) to week 56 was presented based on in-trial data. IWQoL-Lite for CT is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale | 5.4 (18.4) | 4.0 (16.7)

21. Secondary Outcome: Change in IWQoL-Lite for CT: Total Score
Description: Change in IWQoL-Lite for CT total score from baseline (week 0) to week 56 was presented based on in-trial data. IWQoL-Lite for CT is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Score on a scale | 5.7 (17.6) | 4.8 (16.6)

22. Secondary Outcome: Weight Related Sign and Symptom (WRSS) Measure, Categorical Responses
Description: The WRSS measure is a questionnaire under development. The version applied in this study has 10 items that measure the presence and bothersomeness of 10 weight-related symptoms. Each item has a categorical part with answers on the following 5 possible levels: 'Never/Almost never', 'Rarely', 'Sometimes', 'Often' and 'Almost always/Always'. Number of participants in each category at baseline (week 0) and week 56 was presented. Scoring algorithm was not available prior to database lock and therefore it was decided and documented in the statistical analysis plan that WRSS total score was not to be calculated and analyzed.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised participants. "Number analyzed"=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Participants
  Week 0: Joint pain: number analyzed (Participants) | 198 | 196
  Week 0: Joint pain: Almost always/Always | 11 | 5
  Week 0: Joint pain: Never/Almost never | 74 | 85
  Week 0: Joint pain: Often | 17 | 18
  Week 0: Joint pain: Rarely | 47 | 42
  Week 0: Joint pain: Sometimes | 49 | 46
  Week 56: Joint pain: number analyzed (Participants) | 187 | 188
  Week 56: Joint pain: Almost always/Always | 6 | 5
  Week 56: Joint pain: Never/Almost never | 95 | 75
  Week 56: Joint pain: Often | 12 | 17
  Week 56: Joint pain: Rarely | 35 | 39
  Week 56: Joint pain: Sometimes | 39 | 52
  Week 0: Shortness of breath: number analyzed (Participants) | 198 | 196
  Week 0: Shortness of breath: Almost always/Always | 0 | 0
  Week 0: Shortness of breath: Never/Almost never | 131 | 140
  Week 0: Shortness of breath: Often | 3 | 3
  Week 0: Shortness of breath: Rarely | 45 | 32
  Week 0: Shortness of breath: Sometimes | 19 | 21
  Week 56: Shortness of breath: number analyzed (Participants) | 187 | 188
  Week 56: Shortness of breath: Almost always/Always | 1 | 1
  Week 56: Shortness of breath: Never/Almost never | 137 | 111
  Week 56: Shortness of breath: Often | 5 | 3
  Week 56: Shortness of breath: Rarely | 28 | 46
  Week 56: Shortness of breath: Sometimes | 16 | 27
  Week 0: Heat sensitivity: number analyzed (Participants) | 198 | 196
  Week 0: Heat sensitivity: Almost always/Always | 8 | 9
  Week 0: Heat sensitivity: Never/Almost never | 106 | 109
  Week 0: Heat sensitivity: Often | 13 | 16
  Week 0: Heat sensitivity: Rarely | 34 | 31
  Week 0: Heat sensitivity: Sometimes | 37 | 31
  Week 56: Heat sensitivity: number analyzed (Participants) | 187 | 188
  Week 56: Heat sensitivity: Almost always/Always | 2 | 8
  Week 56: Heat sensitivity: Never/Almost never | 92 | 87
  Week 56: Heat sensitivity: Often | 12 | 13
  Week 56: Heat sensitivity: Rarely | 42 | 47
  Week 56: Heat sensitivity: Sometimes | 39 | 33
  Week 0: Sexual desire: number analyzed (Participants) | 198 | 196
  Week 0: Sexual desire: Almost always/Always | 8 | 8
  Week 0: Sexual desire: Never/Almost never | 119 | 121
  Week 0: Sexual desire: Often | 13 | 13
  Week 0: Sexual desire: Rarely | 35 | 32
  Week 0: Sexual desire: Sometimes | 23 | 22
  Week 56: Sexual desire: number analyzed (Participants) | 187 | 188
  Week 56: Sexual desire: Almost always/Always | 6 | 11
  Week 56: Sexual desire: Never/Almost never | 105 | 109
  Week 56: Sexual desire: Often | 18 | 11
  Week 56: Sexual desire: Rarely | 34 | 32
  Week 56: Sexual desire: Sometimes | 24 | 25
  Week 0: Heavy sweating: number analyzed (Participants) | 198 | 196
  Week 0: Heavy sweating: Almost always/Always | 2 | 5
  Week 0: Heavy sweating: Never/Almost never | 101 | 104
  Week 0: Heavy sweating: Often | 15 | 14
  Week 0: Heavy sweating: Rarely | 40 | 38
  Week 0: Heavy sweating: Sometimes | 40 | 35
  Week 56: Heavy sweating: number analyzed (Participants) | 187 | 188
  Week 56: Heavy sweating: Almost always/Always | 1 | 5
  Week 56: Heavy sweating: Never/Almost never | 98 | 92
  Week 56: Heavy sweating: Often | 7 | 16
  Week 56: Heavy sweating: Rarely | 51 | 48
  Week 56: Heavy sweating: Sometimes | 30 | 27
  Week 0: Low physical stamina: number analyzed (Participants) | 198 | 196
  Week 0: Low physical stamina: Almost always/Always | 2 | 8
  Week 0: Low physical stamina: Never/Almost never | 73 | 78
  Week 0: Low physical stamina: Often | 22 | 14
  Week 0: Low physical stamina: Rarely | 56 | 47
  Week 0: Low physical stamina: Sometimes | 45 | 49
  Week 56: Low physical stamina: number analyzed (Participants) | 187 | 188
  Week 56: Low physical stamina: Almost always/Always | 3 | 4
  Week 56: Low physical stamina: Never/Almost never | 77 | 65
  Week 56: Low physical stamina: Often | 15 | 19
  Week 56: Low physical stamina: Rarely | 57 | 56
  Week 56: Low physical stamina: Sometimes | 35 | 44
  Week 0: Foot pain: number analyzed (Participants) | 198 | 196
  Week 0: Foot pain: Almost always/Always | 5 | 7
  Week 0: Foot pain: Never/Almost never | 114 | 108
  Week 0: Foot pain: Often | 17 | 12
  Week 0: Foot pain: Rarely | 34 | 31
  Week 0: Foot pain: Sometimes | 28 | 38
  Week 56: Foot pain: number analyzed (Participants) | 187 | 188
  Week 56: Foot pain: Almost always/Always | 2 | 7
  Week 56: Foot pain: Never/Almost never | 106 | 88
  Week 56: Foot pain: Often | 15 | 14
  Week 56: Foot pain: Rarely | 29 | 39
  Week 56: Foot pain: Sometimes | 35 | 40
  Week 0: Trouble sleeping: number analyzed (Participants) | 198 | 196
  Week 0: Trouble sleeping: Almost always/Always | 6 | 4
  Week 0: Trouble sleeping: Never/Almost never | 119 | 111
  Week 0: Trouble sleeping: Often | 11 | 10
  Week 0: Trouble sleeping: Rarely | 30 | 42
  Week 0: Trouble sleeping: Sometimes | 32 | 29
  Week 56: Trouble sleeping: number analyzed (Participants) | 187 | 188
  Week 56: Trouble sleeping: Almost always/Always | 6 | 3
  Week 56: Trouble sleeping: Never/Almost never | 104 | 98
  Week 56: Trouble sleeping: Often | 15 | 14
  Week 56: Trouble sleeping: Rarely | 38 | 33
  Week 56: Trouble sleeping: Sometimes | 24 | 40
  Week 0: Back pain: number analyzed (Participants) | 198 | 196
  Week 0: Back pain: Almost always/Always | 8 | 6
  Week 0: Back pain: Never/Almost never | 96 | 98
  Week 0: Back pain: Often | 13 | 8
  Week 0: Back pain: Rarely | 49 | 40
  Week 0: Back pain: Sometimes | 32 | 44
  Week 56: Back pain: number analyzed (Participants) | 187 | 188
  Week 56: Back pain: Almost always/Always | 5 | 4
  Week 56: Back pain: Never/Almost never | 93 | 86
  Week 56: Back pain: Often | 13 | 11
  Week 56: Back pain: Rarely | 47 | 45
  Week 56: Back pain: Sometimes | 29 | 42
  Week 0: Low energy: number analyzed (Participants) | 198 | 196
  Week 0: Low energy: Almost always/Always | 0 | 2
  Week 0: Low energy: Never/Almost never | 102 | 90
  Week 0: Low energy: Often | 19 | 12
  Week 0: Low energy: Rarely | 46 | 42
  Week 0: Low energy: Sometimes | 31 | 50
  Week 56: Low energy: number analyzed (Participants) | 187 | 188
  Week 56: Low energy: Almost always/Always | 0 | 4
  Week 56: Low energy: Never/Almost never | 82 | 77
  Week 56: Low energy: Often | 16 | 16
  Week 56: Low energy: Rarely | 49 | 50
  Week 56: Low energy: Sometimes | 40 | 41

23. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c <7% and Weight Loss ≥5%
Description: Percentage of participants who achieved HbA1c <7% and weight loss ≥5% from baseline at week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 39.9 | 13.6

24. Secondary Outcome: Participants Who Achieved (Yes/no): HbA1c <7%, Weight Loss ≥5% and no Documented Symptomatic Hypoglycaemia
Description: Percentage of participants who achieved HbA1c <7%, weight loss ≥5% from baseline and no documented symptomatic hypoglycaemia at week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 10.1 | 3.5

25. Secondary Outcome: Participants Who Achieved (Yes/no): ≥4.3 T-score Points Increase From Baseline in SF-36 Acute Physical Functioning Score
Description: Percentage of participants who achieved ≥4.3 T-score points increase from baseline in SF-36 acute physical functioning score at week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 28.8 | 26.3

26. Secondary Outcome: Participants Who Achieved (Yes/no): ≥3.8 T-score Points Increase From Baseline in SF-36 Acute PCS
Description: Percentage of participants who achieved ≥3.8 T-score points increase from baseline in SF-36 acute PCS at week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 37.9 | 31.3

27. Secondary Outcome: Participants Who Achieved (Yes/no): ≥4.6 T-score Points Increase From Baseline in SF-36 Acute MCS
Description: Percentage of participants who achieved ≥4.6 T-score points increase from baseline in SF-36 acute MCS at week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 14.6 | 11.6

28. Secondary Outcome: Responder Definition Value for IWQoL-Lite for CT Physical Function Domain Score
Description: Percentage of participants who achieve responder definition value for IWQoL-Lite for CT physical function domain score was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 56
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 198 | 198
Percentage of participants | 25.3 | 24.2

29. Secondary Outcome: Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment. Number of AEs from randomisation to until the end of the post-treatment follow-up period (30 days). Results based on in-trial data was presented. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0 to week 56 + 30 days
Population: Safety analysis set (SAS) included all randomised participants exposed to at least one dose of trial drug.
Measure: Number; unit: Adverse events
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Adverse events | 1223 | 1148

30. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0 to week 56 + 30 days
Population: SAS included all randomised participants exposed to at least one dose of trial drug.
Measure: Number; unit: Hypoglycaemic episodes
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Hypoglycaemic episodes | 1538 | 1973

31. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as abdomen; gastrointestinal system; cardiovascular system; central and peripheral nervous system; general appearance; head, eyes, ears, nose, throat (ENT) and neck; lymph node palpation; musculoskeletal system; respiratory system; skin and thyroid gland. The number of participants assessed as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) at baseline (week -1) and week 56 was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week -1, week 56
Population: SAS included all randomised participants exposed to at least one dose of trial drug. "Number analyzed"=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Participants
  Abdomen (week -1) Normal | 165 | 169
  Abdomen (week -1) Abnormal, NCS | 25 | 25
  Abdomen (week -1) Abnormal CS | 5 | 3
  Abdomen (week 56) Normal: number analyzed (Participants) | 185 | 187
  Abdomen (week 56) Normal | 167 | 160
  Abdomen (week 56) Abnormal, NCS: number analyzed (Participants) | 185 | 187
  Abdomen (week 56) Abnormal, NCS | 15 | 24
  Abdomen (week 56) Abnormal, CS: number analyzed (Participants) | 185 | 187
  Abdomen (week 56) Abnormal, CS | 3 | 3
  Gastrointestinal System (week -1) Normal | 185 | 187
  Gastrointestinal System (week -1) Abnormal NCS | 10 | 10
  Gastrointestinal System (week -1) Abnormal CS | 0 | 0
  Gastrointestinal System (week 56) Normal: number analyzed (Participants) | 185 | 185
  Gastrointestinal System (week 56) Normal | 175 | 177
  Gastrointestinal System (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 185
  Gastrointestinal System (week 56) Abnormal NCS | 10 | 8
  Gastrointestinal System (week 56) Abnormal CS: number analyzed (Participants) | 185 | 185
  Gastrointestinal System (week 56) Abnormal CS | 0 | 0
  Cardiovascular System (week-1) Normal | 183 | 182
  Cardiovascular System (week-1) Abnormal NCS | 10 | 15
  Cardiovascular System (week-1) Abnormal CS | 2 | 0
  Cardiovascular System (week 56) Normal: number analyzed (Participants) | 185 | 187
  Cardiovascular System (week 56) Normal | 178 | 175
  Cardiovascular System (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Cardiovascular System (week 56) Abnormal NCS | 6 | 12
  Cardiovascular System (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Cardiovascular System (week 56) Abnormal CS | 1 | 0
  Nervous System (week -1) Normal | 158 | 159
  Nervous System (week -1) Abnormal NCS | 26 | 25
  Nervous System (week -1) Abnormal CS | 11 | 13
  Nervous System (week 56) Normal: number analyzed (Participants) | 185 | 187
  Nervous System (week 56) Normal | 150 | 149
  Nervous System (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Nervous System (week 56) Abnormal NCS | 22 | 24
  Nervous System (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Nervous System (week 56) Abnormal CS | 13 | 14
  General Appearance (week -1) Normal | 150 | 150
  General Appearance (week -1) Abnormal NCS | 39 | 36
  General Appearance (week -1) Abnormal CS | 6 | 11
  General Appearance (week 56) Normal: number analyzed (Participants) | 185 | 187
  General Appearance (week 56) Normal | 156 | 151
  General Appearance (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  General Appearance (week 56) Abnormal NCS | 23 | 27
  General Appearance (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  General Appearance (week 56) Abnormal CS | 6 | 9
  Head, eyes, ENTand Neck (week -1) Normal | 176 | 182
  Head, eyes, ENTand Neck (week -1) Abnormal NCS | 17 | 13
  Head, eyes, ENTand Neck (week -1) Abnormal CS | 2 | 2
  Head, eyes, ENTand Neck (week 56) Normal: number analyzed (Participants) | 185 | 187
  Head, eyes, ENTand Neck (week 56) Normal | 168 | 173
  Head, eyes, ENTand Neck (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Head, eyes, ENTand Neck (week 56) Abnormal NCS | 15 | 12
  Head, eyes, ENTand Neck (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Head, eyes, ENTand Neck (week 56) Abnormal CS | 2 | 2
  Lymph Node Palpation (week -1) Normal | 195 | 197
  Lymph Node Palpation (week -1) Abnormal NCS | 0 | 0
  Lymph Node Palpation (week -1) Abnormal CS | 0 | 0
  Lymph Node Palpation (week 56) Normal: number analyzed (Participants) | 185 | 186
  Lymph Node Palpation (week 56) Normal | 185 | 186
  Lymph Node Palpation (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 186
  Lymph Node Palpation (week 56) Abnormal NCS | 0 | 0
  Lymph Node Palpation (week 56) Abnormal CS: number analyzed (Participants) | 185 | 186
  Lymph Node Palpation (week 56) Abnormal CS | 0 | 0
  Musculoskeletal System (week -1) Normal | 180 | 180
  Musculoskeletal System (week -1) Abnormal NCS | 13 | 16
  Musculoskeletal System (week -1) Abnormal CS | 2 | 1
  Musculoskeletal System (week 56) Normal: number analyzed (Participants) | 185 | 187
  Musculoskeletal System (week 56) Normal | 171 | 171
  Musculoskeletal System (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Musculoskeletal System (week 56) Abnormal NCS | 13 | 14
  Musculoskeletal System (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Musculoskeletal System (week 56) Abnormal CS | 1 | 2
  Respiratory System (week -1) Normal | 192 | 192
  Respiratory System (week -1) Abnormal NCS | 3 | 3
  Respiratory System (week -1) Abnormal CS | 0 | 2
  Respiratory System (week 56) Normal: number analyzed (Participants) | 185 | 187
  Respiratory System (week 56) Normal | 183 | 185
  Respiratory System (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Respiratory System (week 56) Abnormal NCS | 2 | 0
  Respiratory System (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Respiratory System (week 56) Abnormal CS | 0 | 2
  Skin (week -1) Normal | 155 | 156
  Skin (week -1) Abnormal NCS | 36 | 33
  Skin (week -1) Abnormal CS | 4 | 8
  Skin (week 56) Normal: number analyzed (Participants) | 185 | 187
  Skin (week 56) Normal | 150 | 149
  Skin (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Skin (week 56) Abnormal NCS | 28 | 29
  Skin (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Skin (week 56) Abnormal CS | 7 | 9
  Thyroid Gland (week -1) Normal | 183 | 187
  Thyroid Gland (week -1) Abnormal NCS | 10 | 7
  Thyroid Gland (week -1) Abnormal CS | 2 | 3
  Thyroid Gland (week 56) Normal: number analyzed (Participants) | 185 | 187
  Thyroid Gland (week 56) Normal | 180 | 178
  Thyroid Gland (week 56) Abnormal NCS: number analyzed (Participants) | 185 | 187
  Thyroid Gland (week 56) Abnormal NCS | 5 | 6
  Thyroid Gland (week 56) Abnormal CS: number analyzed (Participants) | 185 | 187
  Thyroid Gland (week 56) Abnormal CS | 0 | 3

32. Secondary Outcome: Change in Resting Pulse
Description: Change from baseline (week -1) to week 56 in resting pulse was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week -1, week 56
Population: SAS included all randomised participants exposed to at least one dose of trial drug. "Number analyzed" = participants with available data.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Beats/minute | 2 (9) | -0 (9)

33. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: The ECGs were interpreted by the investigator at baseline (week -1) and week 56 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline and week 56 were presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week -1, week 56
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Participants
  Normal (week -1) | 113 | 133
  Abnormal NCS (week -1) | 78 | 60
  Abnormal CS (week -1) | 4 | 4
  Normal (week 56): number analyzed (Participants) | 185 | 186
  Normal (week 56) | 118 | 126
  Abnormal NCS (week 56): number analyzed (Participants) | 185 | 186
  Abnormal NCS (week 56) | 62 | 57
  Abnormal CS (week 56): number analyzed (Participants) | 185 | 186
  Abnormal CS (week 56) | 5 | 3

34. Secondary Outcome: Change in Laboratory Measurements (Haematology) - Haemoglobin
Description: Change from baseline (week 0) to week 56 in haemoglobin was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
mmol/L | -0.1 (0.5) | -0.1 (0.6)

35. Secondary Outcome: Change in Laboratory Measurements (Haematology) - Haematocrit
Description: Change from baseline (week 0) to week 56 in Haematocrit was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Percentage of red blood cells | -0.4 (2.8) | -0.2 (3.0)

36. Secondary Outcome: Change in Laboratory Measurements (Haematology) - Erythrocytes
Description: Change from baseline (week 0) to week 56 in erythrocytes was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12 cells/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
10^12 cells per liter (10^12 cells/L) | -0.07 (0.27) | -0.04 (0.28)

37. Secondary Outcome: Change in Laboratory Measurements (Haematology) - Thrombocytes, Leukocytes
Description: Change from baseline (week 0) to week 56 in thrombocytes and leukocytes was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
10^9 cells/L
  Thrombocytes: number analyzed (Participants) | 184 | 186
  Thrombocytes | 7 (45) | 7 (46)
  Leukocytes: number analyzed (Participants) | 185 | 186
  Leukocytes | -0.22 (1.41) | -0.24 (1.28)

38. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Albumin
Description: Change from baseline (week 0) to week 56 in albumin was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Grams per deciliter (g/dL) | -0.1 (0.2) | -0.1 (0.2)

39. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Alkaline Phosphatase, Alanine Aminotransferase, Amylase, Aspartate Aminotransferase and Lipase
Description: Change from baseline (week 0) to week 56 in alkaline phosphatase, alanine aminotransferase, amylase, aspartate aminotransferase and lipase was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Units per liter (U/L)
  Alkaline Phosphatase: number analyzed (Participants) | 185 | 189
  Alkaline Phosphatase | -1 (16) | -0 (15)
  Alanine Aminotransferase: number analyzed (Participants) | 185 | 188
  Alanine Aminotransferase | -5 (15) | -6 (18)
  Amylase: number analyzed (Participants) | 185 | 189
  Amylase | 13 (73) | -1 (22)
  Aspartate aminotransferase: number analyzed (Participants) | 185 | 189
  Aspartate aminotransferase | -3 (11) | -3 (14)
  Lipase: number analyzed (Participants) | 185 | 189
  Lipase | 30 (143) | -8 (47)

40. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Bicarbonate, Total Calcium, Potassium, Sodium and Urea
Description: Change from baseline (week 0) to week 56 in bicarbonate, total calcium, potassium, sodium and urea was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
mmol/L
  Bicarbonate serum: number analyzed (Participants) | 156 | 171
  Bicarbonate serum | 0 (2) | -0 (2)
  Total Calcium: number analyzed (Participants) | 185 | 189
  Total Calcium | -0.00 (0.11) | -0.02 (0.14)
  Potassium: number analyzed (Participants) | 185 | 189
  Potassium | -0.0 (0.5) | -0.0 (0.5)
  Sodium: number analyzed (Participants) | 185 | 189
  Sodium | -1 (2) | -0 (3)
  Urea: number analyzed (Participants) | 185 | 189
  Urea | 0.1 (1.5) | 0.1 (1.4)

41. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Total Bilirubin and Creatinine
Description: Change from baseline (week 0) to week 56 in total bilirubin and creatinine was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Micromoles per liter (umol/L)
  Total Bilirubin: number analyzed (Participants) | 185 | 188
  Total Bilirubin | 1.0 (3.9) | 0.6 (3.6)
  Creatinine: number analyzed (Participants) | 185 | 189
  Creatinine | -0.1 (8.7) | -0.2 (8.4)

42. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - High Sensitive C-reactive Protein
Description: Change from baseline (week 0) to week 56 in high sensitive C-reactive protein was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Milligrams per liter (mg/L) | -1.40 (8.02) | -1.29 (10.07)

43. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - eGFR
Description: Change from baseline (week 0) to week 56 in estimated GFR serum using Modification of Diet in Renal Disease (MDRD) formula was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Milliliters per minute per 1.73m^2
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Milliliters per minute per 1.73m^2 | 0 (13) | 1 (13)

44. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Uric Acid
Description: Change from baseline (week 0) to week 56 in uric acid was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
mg/dL | -0.2 (1.0) | -0.0 (0.9)

45. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Calcitonin
Description: Change from baseline (week 0) to week 56 in calcitonin was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Nanograms per liter (ng/L) | 0.0 (1.5) | 0.0 (1.4)

46. Secondary Outcome: Change in Laboratory Parameters (Biochemistry) - Thyroid Stimulating Hormone
Description: Change from baseline (week 0) to week 56 in thyroid stimulating hormone was presented based on in-trial data. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact.
Time Frame: Week 0, week 56
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Milli-international units per liter
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 195 | 197
Milli-international units per liter | -0.0842 (1.2233) | 0.1002 (0.9493)

ADVERSE EVENTS:
Time Frame: From the date of first dose of trial product (week 0) to end of treatment (week 56) + post treatment follow-up of 30 days.
Description: Evaluation of safety was based on SAS which comprised of all randomised participants who received at least one dose of trial product.
  AEs with onset during the on-treatment observation period (the period when participants were exposed to trial product) were considered treatment-emergent.
Arm/Group | Liraglutide 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/197
Serious Adverse Events (participants affected / at risk) | 16/195 | 19/197
Other Adverse Events (participants affected / at risk) | 162/195 | 141/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=195) | Placebo (N=197)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metaphyseal corner fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=195) | Placebo (N=197)
Abdominal discomfort (Gastrointestinal disorders) | 11 (17) | 8 (11)
Abdominal pain upper (Gastrointestinal disorders) | 12 (17) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 24 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (17)
Constipation (Gastrointestinal disorders) | 28 (36) | 17 (21)
Decreased appetite (Metabolism and nutrition disorders) | 19 (24) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 45 (77) | 30 (54)
Dizziness (Nervous system disorders) | 13 (18) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 12 (13) | 5 (5)
Fatigue (General disorders) | 14 (18) | 10 (11)
Gastroenteritis (Infections and infestations) | 15 (15) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (12) | 2 (2)
Headache (Nervous system disorders) | 29 (36) | 29 (47)
Hypertension (Vascular disorders) | 4 (4) | 12 (14)
Influenza (Infections and infestations) | 12 (14) | 22 (26)
Nasopharyngitis (Infections and infestations) | 42 (48) | 36 (49)
Nausea (Gastrointestinal disorders) | 58 (105) | 23 (27)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (12)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (9) | 12 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (17) | 19 (21)
Sinusitis (Infections and infestations) | 9 (11) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 24 (32) | 29 (37)
Urinary tract infection (Infections and infestations) | 7 (12) | 19 (22)
Vomiting (Gastrointestinal disorders) | 32 (53) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT02963922/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT02963922/SAP_001.pdf